CLINICAL TRIAL: NCT06700434
Title: Clinical Evaluation of In-office Bleaching With Low, Medium, and High Concentrate Hydrogen Peroxide: A 6-month a Double-blinded Randomized Controlled Trial
Brief Title: Clinical Efficacy of In-office Bleaching With Different Concentrations of Hydrogen Peroxide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Hanife ALTINIŞIK, Associate Professor, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TGA-2023-8355
Record Dates: First submitted 2024-11-15; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-03

CONDITIONS: Tooth Discoloration
Keywords: Hydrogen Peroxide; In-office bleaching; Randomized clinical trial; Tooth sensitivity; Whitening effectiveness; Quality of life
MeSH Terms: conditions — Tooth Discoloration; Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: A 6-month a double-blinded randomized controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Inclusion criteria: Females and males (least 18 years old), good oral and general health, no periodontal disease, no caries, and teeth colored A3 or darker according to the VITA Easy Shade Guide (VITA Zanhnfabrik, BadSckingrn, Germany).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HP18 (Active Comparator): Bleaching agent containing Hydrogen Peroxide 18% and nano- hydroxyapatite
  Interventions: Other: Bleaching treatment
- HP25 (Active Comparator): Bleaching agent containing Hydrogen Peroxide 20% and nano- hydroxyapatite
  Interventions: Other: Bleaching treatment
- HP40 (Active Comparator): Bleaching agent containing Hydrogen Peroxide 40% and nano- hydroxyapatite
  Interventions: Other: Bleaching treatment

INTERVENTIONS:
Other: Bleaching treatment — After the lip retractor (OptraGate, Ivoclar Vivadent, Schaan, Liechtenstein) was placed, the gingival barrier protection (Biowhiten, Biodent Ltd., İstanbul, Turkey) included in the products was applied to the upper and lower arches from premolar to premolar at the beginning of each session and removed after each treatment. The bleaching gels were applied according to the manufacturer and removed after the recommended period with a disposable surgical saliva ejector, cleaned with gauze and washed with air-water spray. Two bleaching sessions were performed at a 1-week interval. Participants were advised to maintain regular oral hygiene by brushing with toothpaste that does not contain desensitizing or whitening ingredients.
  HP18 is applied in 5 applications of 10 minutes per session. HP25 is applied in 3 applications of 15 minutes per session. HP40 is applied in 3 applications of 15 minutes per session.

SUMMARY:
Objective: The study evaluated the longevity, effectiveness, sensitivity and impact on the oral health-related quality of life of in-office dental bleaching using low, medium, and high concentrate hydrogen peroxide.

Material and Methods: Randomized, parallel, and double-blinded clinical trial was performed with 54 participants using18% hydrogen peroxide (HP), 20%HP, and 40%HP in-office bleaching agent. Tooth color was evaluated at baseline, after the 1st session bleaching, after the 2st session bleaching and 6 months (T5) after finishing the bleaching using spectrophotometer. Tooth sensitivity was measured with the Visual Analog Scale at baseline, immediately after bleaching, after 1 day, and after 7 days. The impact on quality of life was evaluated using the Oral Health Impact Profile (OHIP) questionnaire at baseline, and 6 months after bleaching.

ELIGIBILITY:
Inclusion Criteria:

* Women and men (at least 18 years old)
* People with good oral and general health
* People without periodontal disease
* Teeth without caries
* Teeth A3 or darker according to the VITA Easy Shade Guide (VITA Zanhnfabrik, BadSckingrn, Germany)

Exclusion Criteria:

* Having undergone teeth bleaching procedure in the last 2 years,
* People with tooth sensitivity,
* Use of fixed orthodontic appliances or prostheses on upper and/or lower anterior teeth,
* People with gingival recession,
* Discoloration due to parafunction, tetracycline or fluorosis,
* Smokers,
* Tooth fracture.

Ages: 21 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Tooth Shade evaluation | baseline, immediately after the first bleaching session, immediately after the second whitening session (7 days after the first bleaching), 180 days after the first bleaching session
  Tooth color was objectively evaluated using VitaTM Easy Shade V spectrophotometer (VITA Zanhnfabrik, BadSckingrn, Germany). The assesment was performed with daylight (10 a.m.to 2 p.m.) considering a 6 mm area situated in the middle section of the labial surface of the upper central incisors. In order to ensure consistency, alginate impressions were taken of the upper dental arches of each participant and stone molds were created. The custom trays were fabricated by using a 2mm Essix plate (Essix C; Dentsply, FL, USA) in a vacuum press machine (Ministar, Scheu, Iserlohn, Nordrhein-Westfalen Germany). 6 mm wide holes were drilled in the middle third of the buccal face of the central incisors on this trays to serve as a guide for using Easyshade V.

SECONDARY OUTCOMES:
Tooth sensitivity evaluation | baseline, immediately after the first bleaching session, two hours later, and 7 days later.
  To measure tooth sensitivity, participants indicated their discomfort level using a Visual Analog Scale (VAS).23 This scale is represented by a horizontal line measuring 10 centimeters in length. The endpoint of the line labeled "no pain" represents the absence of discomfort, while the opposite endpoint labeled "worst pain" represents the highest level of discomfort.

OTHER OUTCOMES:
Impact of oral condition on quality of life | baseline and 180 days after bleaching
  The OHIP-14 questionnaire was utilized to evaluate the quality of life.24 This questionnaire consists of seven different domains and a total of 14 questions aimed at assessing one's quality of life. Responses to questions were determined by selecting one choice from a Likert scale. The scale included options like never (0 points), rarely (1 points), sometimes (2 points), often (3 points), and always (4 points), each corresponding to a certain number of points. A person's oral health-related quality of life (OHRQoL) is negatively affected when the average value of seven dimensions is higher.

CONTACTS AND LOCATIONS:
Overall Officials: Associate Prof, Study Director — Gazi University; Research assistant, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altinisik H, Nezir M. Clinical evaluation of in-office bleaching with low, medium, and high concentrate hydrogen peroxide: a 6-month a double-blinded randomized controlled trial. Clin Oral Investig. 2025 Apr 21;29(5):260. doi: 10.1007/s00784-025-06348-8. PMID 40259078